CLINICAL TRIAL: NCT04041557
Title: Intellectual and Executive Functions in Relation to Cerebral MRI in Young Adults With Congenital Heart Disease
Brief Title: Executive Functions in Adults With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Bea Latal, Prof. Bea Latal, University Children's Hospital, Zurich
Other Study IDs: GUCHZurich
Record Dates: First submitted 2019-07-04; First posted 2019-08-01 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adults with CHD: Adults with congenital heart disease 18-32 years of age
- controls: healthy peers

SUMMARY:
Research in children with congenital heart disease (CHD) requiring cardiopulmonary bypass surgery in the neonatal period or during early childhood has shown that the survival rate for this population has dramatically increased, also for those with the most severe forms of CHD. However, they are at significant risk for neurodevelopmental impairments, persisting into adolescence. Our research group showed that adolescents with CHD have smaller brain volumes than controls and that volume reduction correlates with poorer neurocognitive functioning. It is not known whether similar changes can also be found in adults with CHD (ACHD).

Aims:

1. To determine intellectual and executive functions in young adults with congenital heart disease after childhood cardiopulmonary bypass surgery and to relate these findings to results on cerebral magnetic resonance imaging (MRI).
2. To evaluate risk factors for adverse outcome and alteration on cerebral MRI.
3. To examine the effect of poorer intellectual and executive functioning on academic achievement, quality of life, and psychosocial functioning.

Methodology:

Outcome variables: Intellectual and executive functioning as well as cerebral MRI.

Participants: Study subjects will be recruited from a large cohort that has been enrolled in a study on quality of life in ACHD. The investigators aim to include a maximum of 60 subjects per group (ACHD, controls). Variables and risk factors influencing outcome have already been assessed through that study. Cerebral MRI will be analysed for structural abnormalities, and volumetric, morphometric as well as connectivity analyses will be performed to comprehensively characterize cerebral architecture in ACHD and to compare it with that of healthy controls.

Inclusion criteria: Patients with congenital heart disease, cardiopulmonary bypass surgery during childhood, age 18 to 30 years Exclusion criteria: Known genetic syndromes or chromosomal abnormalities as well as other congenital or acquired diseases leading to mental disabilities, exclusion criteria for cerebral MRI.

DETAILED DESCRIPTION:
The overall aim of our project is to study intellectual and executive functions in relation to cerebral magnetic resonance imaging (MRI) in young adults with severe congenital heart disease (CHD). Risk factors for poorer function and altered brain structure will be examined. This will extend the knowledge on the spectrum of potential long-term impairments, risk factors and the effect on the patient's quality of life. Only a better understanding of the spectrum and contributing factors of neurocognitive impairments in adults will allow for an early therapy in childhood and will prevent or ameliorate long-term sequelae for patients with CHD.

Specific aims:

1. To determine the intellectual and executive function of young adults with congenital heart disease after cardiopulmonary bypass surgery during infancy or childhood Hypothesis: Intellectual outcome is within the normal range but below that of controls and assume to find specific difficulties in certain areas of executive functions.
2. To perform cerebral MRI and perform morphometric analyses Hypothesis: Cerebral volumes will be smaller and regional white matter microstructure will be altered, which correlate with intellectual and executive function
3. To determine patient and medical risk factors associated with adverse outcome Hypothesis: Disease severity correlates with intellectual outcome.
4. To determine the associations between intellectual and executive function and quality of life Hypothesis: Functional outcome correlates with quality of life.

Subjects:

The patients and controls have participated in a study on quality of life in adults with CHD and will be asked to return for this part of the study. So far, 180 patients and 145 controls have been enrolled.

Inclusion Criteria:

* Patients with congenital heart disease
* Bypass surgery for congenital heart disease
* Male and female subject 18 to 30 years of age
* Written informed consent by the participant after information about the project
* In command of the German language
* No exclusion criteria for cerebral MRI

Exclusion Criteria:

* Known genetic syndromes or chromosomal abnormalities as well as other congenital or acquired diseases leading to mental disabilities
* Exclusion criteria for cerebral MRI

Outcome measures:

Intelligence will be assessed with the Wechsler Adult Intelligence Scale IV edition.

A large battery using standardized tests will be administered for the executive function assessment. This includes the following domains: Working and visual memory, inhibition, flexibility, planning, fluency, attention and questionnaires will assess the everyday functioning regarding executive functions (behavior rating inventory of executive functions-BRIEF).

Medical and sociodemographic data These data have already been obtained by the ongoing study.

Cerebral MRI MRI will be performed with a 3.0-T whole-body system (Signa Twinspeed Excite; GE Healthcare, Milwaukee, Wisconsin). Three-dimensional anatomic images of the entire brain will be obtained using a T1-weighted gradient echo pulse sequence (repetition time, 25 msec; echo time, 5 msec) and a T2-weighted spin echo pulse sequence (repetition time,6660 msec; echo time, 97.6 msec).

Time schedule Recruitment and testing phase 6-9 months, data entry, data control and preliminary data analysis 3 months.

Start of the project: January 1st, 2017, duration: 1 year.

Statistical Plan The sample size estimated is 51 participants per group given a two-sided alpha of 0.05 and a power of 90% resulting in a total of 102 participants for the study. In order to control for drop-outs, each group will comprise 60 subjects. Data will be analyzed using SPSS statistic software version 23 (SPSS inc., Chicago). Parametric or non-parametric procedures will be used to compare patients and controls with regard to outcome variables. To examine the role of predictors for the outcomes multivariate regression analyses will be performed.

Ethics Ethical approval is available for the assessment of neurocognitive and executive functions. An amendment is currently being submitted for the cerebral MRI part.

ELIGIBILITY:
Inclusion Criteria:

•Congenital heart disease

Exclusion Criteria:

•Genetic condition

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: adults with congenital heart disease followed at the University Hospital Zürich
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Intellectual performance | 1.1.17-30.9.18
  short version of the adult WISC form
Executive function global score | 1.1.17-30.9.18
  A score that is derived from averaging the T-values of the following executive function tests: color-word-interference test of the Delis-Kaplan-Executive Function System (D-KEFS) and the stop-signal task of the STOP-IT-both measuring inhibition, the S word of the Regensburger Wortflüssigkeitstest-measuring fluency, the Standardized Links' Probe-measuring planning, and the Trail Making Test -measuring cognitive flexibility.
  Value: Mean 50 (+/-10), higher value better performance

SECONDARY OUTCOMES:
total brain volume on cerebral MRI | 1.1.17-30.9.18
  the total brain volume will be measured with a standardized protocol (free surfer) and expressed as mm3 (larger number equals larger brain)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kessler N, Feldmann M, Schlosser L, Rometsch S, Brugger P, Kottke R, Knirsch W, Oxenius A, Greutmann M, Latal B. Structural brain abnormalities in adults with congenital heart disease: Prevalence and association with estimated intelligence quotient. Int J Cardiol. 2020 May 1;306:61-66. doi: 10.1016/j.ijcard.2020.02.061. Epub 2020 Feb 24. PMID 32143921